CLINICAL TRIAL: NCT01428947
Title: Study of Cognitive Function Before and After Coronary Angiography
Brief Title: Does Coronary Angiography Cause Cognitive Dysfunction?
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Tornvall, Docent, Karolinska Institutet
Other Study IDs: KI-angio-2
Record Dates: First submitted 2011-08-26; First posted 2011-09-05 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Heart Disease; Heart Valve Diseases
MeSH Terms: conditions — Coronary Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary angiography: Patents scheduled for elective coronary angiography
  Interventions: Procedure: Arterial approach

INTERVENTIONS:
Procedure: Arterial approach — Randomization to right radial or femoral approach
  Other Names: Coronary arteriography

SUMMARY:
The purpose of the study is to study if coronary angiography cause cognitive dysfunction.

DETAILED DESCRIPTION:
We have previously shown, using transcranial doppler, that coronary angiography cause cerebral microembolism. Cerebral microemboli were more common using the radial than femoral approach. Previously, cerebral microembolism has been associated with new cerebral lesions on MRI. The clinical significance of these new lesions is not determined. The primary aim of this pilot study is to see if coronary angiography cause cognitive dysfunction determined by the MoCA-test. A secondary aim is to relate cognitive dysfunction to cerebral microembolism measured by transcranial doppler. A third aim is to study potential differences between the femoral and radial approaches.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary angiography irrespective of cause

Exclusion Criteria:

* Previous CABG, language problems, not willing to participate

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective coronary angiography at one center
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in cognitive dysfunction from baseline to two days after coronary angiography | Baseline and two days
  The Montreal Cognitive Assesment test will be performed before, 2 and 30 days after coronary angiography

SECONDARY OUTCOMES:
Number of patients with cerebral microemboli | Baseline
  Cerebral microembolism will be studied by transcraniell doppler at the time of angiography. Findings will be related to change in cognitive function between baseline and two days.

CONTACTS AND LOCATIONS:
Overall Officials: Per - Tornvall, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Cardiology Clinic, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Jurga J, Nyman J, Tornvall P, Mannila MN, Svenarud P, van der Linden J, Sarkar N. Cerebral microembolism during coronary angiography: a randomized comparison between femoral and radial arterial access. Stroke. 2011 May;42(5):1475-7. doi: 10.1161/STROKEAHA.110.608638. Epub 2011 Mar 10. PMID 21393589